CLINICAL TRIAL: NCT00003568
Title: A Randomized Phase II Trial of a Mutated gp100 Melanoma Peptide (g209-217(210M) With Hight Dose Interleukin-2 (IL-2) in HLA-A2.1+Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy With High-Dose Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CWG-UIC-T98-0027; CDR0000066634 (Registry Identifier: PDQ (Physician Data Query)); NCI-T98-0027
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2005-11

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response that will kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells.

PURPOSE: Randomized phase II trial to study the effectiveness of vaccine therapy with interleukin-2 in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the antitumor activity of gp100:209-217 (210M), a melanoma peptide derived from gp100 mixed with Montanide ISA-51, in combination with high-dose interleukin-2 (IL-2) administered by various schedules in patients with advanced melanoma.
* Examine the effect of the addition of gp100:209-217 (210M) peptide vaccine to high-dose IL-2 on the toxicity of the treatment in these patients.
* Define the induction of T-cell responses to gp100:209-217 (210M) peptide and its gp100 (parent) protein by ELISA with interferon gamma production or CTL precursor frequencies in these patients after the initial course of treatment.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior therapy (adjuvant interferon vs chemotherapy for advanced disease vs both vs none), ECOG performance status (0 vs 1), and number of organ sites involved (1 vs more than 1). Patients are randomized into 1 of 3 treatment arms. (Arm III closed to accrual as of 11/30/1998.)

* Arm I: Patients receive vaccination comprising gp100:209-217 (210M) peptide mixed with Montanide ISA-51 subcutaneously on days 1, 22, 43, and 64. Patients also receive high-dose interleukin-2 (IL-2) IV over 15 minutes every 8 hours on days 2-6 and 16-20.
* Arm II: Patients receive vaccination as in arm I on days 1, 22, 43, and 64. Patients also receive high-dose IL-2 as in arm I on days 44-48 and 60-64. Patients who demonstrate rapid visible disease progression during the initial 4 weeks of therapy while maintaining good performance status may begin high-dose IL-2 on day 23.
* Arm III (closed to accrual as of 11/30/1998): Patients receive vaccination as in arm I on day 1 and then high-dose IL-2 as in arm I on day 2. Patients with nonhematologic toxicity may only receive vaccination on weeks 4, 7, and 10. Other patients may also receive IL-2 beginning on day 2 of each treatment week (4, 7, and 10) for up to 14 doses.

Patients in each arm may receive up to a total of 3 courses of treatment.

Patients are followed until death.

PROJECTED ACCRUAL: Approximately 90 patients (25 patients for arms I and II and 40 patients for arm III [arm III closed to accrual as of 11/30/1998]) will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed clearly progressive metastatic or unresectable melanoma
* Must be HLA-A2.1 positive
* Measurable disease
* No active brain metastases, leptomeningeal disease, or seizure disorder

  * More than 4 months since prior definitive therapy (surgery or radiotherapy) for brain metastases and must not have evidence of disease on brain CT scan or MRI
* No ascites or pleural effusions

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1 OR
* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No congestive heart failure
* No symptoms of coronary artery disease
* No serious cardiac arrhythmias
* No evidence of prior myocardial infarction on EKG
* Normal cardiac stress test required for all patients over 40 years

Pulmonary:

* FEV_1 greater than 2.0 liters or at least 75% of predicted
* No chronic obstructive pulmonary disease

Other:

* HIV negative
* No significant systemic infection
* No contraindication to use of pressor agents
* No history of major psychiatric illness
* No other major illness that would significantly increase the risk of immunotherapy
* No other active malignancy except surgically cured nonmelanoma skin cancer or carcinoma in situ or stage I carcinoma of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interleukin-2
* At least 4 weeks since prior vaccine therapy or other cytokine therapy

Chemotherapy:

* One prior chemotherapy regimen allowed
* At least 4 weeks since prior chemotherapy (6 weeks for carmustine or lomustine) and recovered

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to areas of measurable disease unless there has been clearly progressive disease in this site or there is measurable disease outside of areas of prior radiation
* At least 2 weeks since prior radiotherapy for local control or palliative therapy and recovered

Surgery:

* See Disease Characteristics
* Recovered from prior major surgery
* No prior organ allografts

Other:

* No antihypertensive therapy within 24 hours prior to interleukin-2

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-11; Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Gustin, MD, Study Chair — University of Illinois at Chicago
Locations (9):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Center at Our Lady of Mercy Medical CenterOur, The Bronx, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas